CLINICAL TRIAL: NCT04192006
Title: A Prospective Randomised Controlled Trial Comparing the Biochemical, Thermal, and Macroscopic Soft Tissue Outcomes in Conventional Jig-based Total Knee Arthroplasty Versus Mako Robotic-arm Assisted Total Knee Arthroplasty
Brief Title: Inflammatory Response Conventional Total Knee Replacement Versus Mako Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Stryker EU Operations BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17/0742
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis; Arthritis; Surgery
Keywords: biomechanical; inflammation; mako robot; makoplasty; soft tissue injury; total knee arthroplasty; total knee replacement; thermal
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis; Inflammation; Soft Tissue Injuries | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional (Active Comparator): Jig-based procedure
  Interventions: Device: Total Knee Arthroplasty
- Robotic arm-assist (Experimental): Mako robotic-arm assist based procedure
  Interventions: Device: Total Knee Arthroplasty

INTERVENTIONS:
Device: Total Knee Arthroplasty — Surgical implantation of prosthetic knee using robotic-arm assist

SUMMARY:
Total knee Arthroplasty (TKA) is a highly effective treatment for knee osteoarthritis. Mid- to long-term follow-up studies have shown good clinical outcomes following TKA; despite these results, there is a high incidence of patient dissatisfaction; 20% of patients reporting dissatisfaction in otherwise uncomplicated procedures.

One reason for early dissatisfaction may be the trauma of surgery may lead to localised and systemic inflammatory responses that impair postoperative clinical recovery; this in turn influences long-term functional outcomes. Surgical techniques that limit the insult of surgery and help to restore the patient's native knee anatomy and kinematics may help to improve clinical outcomes, functional recovery, and patient satisfaction.

The technical objectives of surgery are to restore limb alignment, preserve the joint line, balance flexion and extension gaps, and maintain the normal Q angle for optimal patella tracking. Compromise to the periarticular soft tissue structures may compromise postoperative clinical and functional recovery, reduce stability, and decrease implant survivorship. In conventional jig-based (CO) TKA, bone cuts are most commonly performed using measured resection or gap balancing. The manual error associated with inadvertent soft tissue release during preparation for implantation or tissue damage from the saw blades is an accepted part of the procedure.

The evolution of surgical technology has led to the development of robotic-arm assisted TKA, which uses three dimensional images of the patient's native knee anatomy to guide bone resection and optimise implant positioning. The second-generation RIO Robotic Arm Interactive Orthopaedic system (Mako surgical) uses preoperative computerised tomography scans to build a computer-aided design (CAD) model of the patient's knee joint. The Mako robotic software processes this information to calculate the volume of bone requiring resection and creates a three-dimensional haptic window for the RIO robotic arm to resect.

In short, the robotic technology in TKA allows execution of the preoperative surgical plan without undue soft tissue release, inadvertent trauma from power tools, and minimal trauma to bone surfaces. Conceptually, this Mako TKA should have reduced soft tissue trauma and inflammatory response as assessed with inflammatory cytokines compared to CO TKA.

The overall aim of this single centre, prospective randomised controlled trial is to determine differences in the inflammatory response between CO TKA and Mako TKA.

A comprehensive range of local and systemic biochemical markers, thermal response, and macroscopic soft tissue injury outcomes between the two groups will be recorded and correlated to clinical and functional outcomes over 2-year postoperative. Patients undergoing CO TKA will form the control group and those undergoing Mako TKA will form the investigation group.

ELIGIBILITY:
Inclusion Criteria:

* Patient has symptomatic knee osteoarthritis requiring primary TKA
* Patient and surgeon are in agreement that TKA is the most appropriate treatment
* Patient is fit for surgical intervention following review by surgeon and anaesthetist
* Patient is between 18-80 years of age at time of surgery
* Gender: male and female
* Patient must be capable of giving informed consent and agree to comply with the postoperative review program
* Patient must be a permanent resident in an area accessible to the study site
* Patient must have sufficient postoperative mobility to attend follow-up clinics and allow for radiographs to be taken

Exclusion Criteria:

* Patient is not suitable for routine primary TKA e.g. patient has ligament deficiency that requires a constrained prosthesis
* Patient has inflammatory arthritis e.g. Rheumatoid arthritis
* Patient has local or systemic autoimmune disease
* Past medical history of cancer or chronic illness
* Patient has symptomatic arthritis of the contralateral knee

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Serum CRP level | 48 hours post-op
  Serum CRP level

SECONDARY OUTCOMES:
C-reactive Protein (CRP) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Interleukin-1 beta (IL1 beta) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Interleukin-6 (IL6) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Tumour necrosis Factor alpha (TNFalpha), | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Creatine Kinase (CK) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Creatine Phosphokinase (CPK) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Full blood count (FBC) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Erythrocyte sedimentation rate (ESR) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Myoglobin (MG) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Lactate dehydrogenase (LDH) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
Urea and Electrolytes (U&Es) | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days following TKA
  Systemic inflammation as assessed by the serial measurement of serum inflammatory cytokines and enzyme markers of soft tissue injury
IL-6 | 6 and 24 hours following surgery
  Local inflammatory response as assessed using intraarticular drain fluid
Interleukin-8 (IL-8) | 6 and 24 hours following surgery
  Local inflammatory response as assessed using intraarticular drain fluid
TNFalpha | 6 and 24 hours following surgery
  Local inflammatory response as assessed using intraarticular drain fluid
Thermal response to inflammation | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days.
  skin temperature over the operated knee joint preoperatively and postoperatively
Soft tissue injury prior to implantation of femoral and tibial prostheses | 28 days post op
  macroscopic examination of the periarticular soft tissues
Operating time | 28 days post op
  Operating time (minutes).
Time to discharge | 28 days post op
  Time to discharge (hours).
Pain in knee | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days
  Subjective score. Pain as assessed using the Visual analogue score (VAS) following surgery. Patient uses line delineated at left hand end with '0' and '10' at the right hand end. 0= no pain; 10 = the most pain. Patient indicates where they feel their pain fits onto this score.
Analgesia requirements | 6 hours, 1 day, 2 days, 3 days, 7 days, and 28 days.
  Analgesia requirements following surgery
Oxford knee score (OKS) | Pre-op; 4 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. 48 is best score and 0 worst score
Short form health survey of 12 items (SF-12) | Pre-op; 4 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure. Questions concerning attitudes to physical and mental heath with 12 questions combined to give overall norm-based values; higher score better, lower score worse.
Knee injury and osteoarthritis outcome score (KOOS) | Pre-op; 4 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire. 6 separate domains including pain, stiffness, quality of life, symptoms, and function; each domain creates percentage with overall cumulative percentage achieved; best score 100%
Western Ontario and Mcmaster Universities Arthritis Index (WOMAC) | Pre-op; 4 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome questionnaire evaluating pain, stiffness and disability in affected joint
European Quality of Life questionnaire with 5 dimensions for adults (EQ-5D) | Pre-op; 4 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure with 5 domains; score -1 to 1, with 1 being best score

CONTACTS AND LOCATIONS:
Overall Officials: Fares S Haddad, Study Chair — UCL Hospitals NHS Foundation Trust
Locations (1):
- University College London Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan